CLINICAL TRIAL: NCT03039569
Title: Assessing Home Food Environment and Diabetes Self-management Among Adult Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16200
Record Dates: First submitted 2017-01-24; First posted 2017-02-01 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes patients; Diabetes self-management; Cardiovascular diseases awareness; Home food environment; Text message
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text messaging (Experimental): Participants will receive 3 messages weekly consisting of nutrition education and diabetes self-management information and skills for 3 months (12 weeks).
  Interventions: Behavioral: Text messaging
- Control (No Intervention): Participants will not receive text message intervention. This is the measurement-only group

INTERVENTIONS:
Behavioral: Text messaging — The messages will consist of information on how to increase fruits and vegetables and reduce high-fat and sugary foods intake, increase the availability of fruits and vegetables and reduce high-fat and sugary foods in the home, strategies to increase diabetes self-management skills, and awareness of cardiovascular disease risk perception and knowledge. The text messages will be derived from the American Association of Diabetes Educator (AADE) handouts ("Reducing Risks", "Monitoring", "Healthy Coping", "Problem Solving", "Taking Medication", "Healthy Eating", and "Exercise"). The control group will not receive text messages
  Arms: Text messaging

SUMMARY:
In this project the investigators examined the impact of diabetes self-management education using text messaging on increasing awareness of CVD risk perception, dietary intake, physical activity, and diabetes self-management among adults with type 2 diabetes using a quasi experimental design. The study sample included 79 adult type 2 diabetes patients (30 years or older). The recruited adult type 2 diabetes patients were assigned into the intervention group (40 participants) and control group (39 participants). The intervention group received 3 messages weekly consisting of nutrition education and diabetes self-management information and skills for 3 months (12 weeks). The messages consisted of information on how to increase fruits and vegetables and reduce high-fat and sugary foods intake, increase the availability of fruits and vegetables and reduce high-fat and sugary foods in the home, strategies to increase diabetes self-management skills, and awareness of cardiovascular disease risk perception and knowledge. The text messages were derived from the American Association of Diabetes Educator (AADE) handouts ("Reducing Risks", "Monitoring", "Healthy Coping", "Problem Solving", "Taking Medication", "Healthy Eating", and "Exercise") Text messages were positive and motivating and included a link to a specific AADE7 handout that allows participants to open and retrieve the specific AADE7 handout. The control group did not receive text messages. The participants (both intervention and control group) completed surveys at baseline (before study begins) and at the conclusion of the study (at three month of the intervention) about their dietary and lifestyle habits, diabetes self-care management activities, and awareness of cardiovascular diseases. We collected also collect patient's self-report Hemoglobin A1C values at baseline and at the conclusion of the study (at three month of the intervention).

DETAILED DESCRIPTION:
Type 2 diabetes and its complications have become an important public health problem, affecting nearly 350 million adults worldwide. However, successfully managing type 2 diabetes through proper nutrition and healthy lifestyles remains challenging for many diabetes patients. In this proposed project the investigators examined the impact of diabetes self-management education using text messaging on increasing awareness of CVD risk perception, dietary intake, physical activity, and diabetes self-management, and quality of life among adults with type 2 diabetes among adults with Type 2 diabetes using a quasi experimental design. The study sample included 79 adult type 2 diabetes patients (30 years or older). Inclusion criteria for the study sample of adult type II diabetes patients were: adults ages 30 or older, English speaking, and Hemoglobin A1C levels > 6.5%.

Adult type 2 diabetes patients were recruited from the Center for Diabetes & Nutritional Health, an outpatient diabetes clinic of Methodist Hospital in Omaha with the assistance of Certified Diabetes Educators and Registered Dietitians. Diagnosis of type 2 diabetes were based on patient self-report and verified by the Co-Primary Investigator (who is Certified Diabetes educator and registered dietitian at the Methodist Hospital. The recruited adult type 2 diabetes patients were assigned into the intervention group (40 participants) and control group (39 participants). The intervention group received 3 messages weekly consisting of nutrition education and diabetes self-management information and skills for 3 months (12 weeks). The messages consisted of information on how to increase fruits and vegetables and reduce high-fat and sugary foods intake, increase the availability of fruits and vegetables and reduce high-fat and sugary foods in the home, strategies to increase diabetes self-management skills, and awareness of cardiovascular disease risk perception and knowledge. The text messages were derived from the American Association of Diabetes Educator (AADE) handouts ("Reducing Risks", "Monitoring", "Healthy Coping", "Problem Solving", "Taking Medication", "Healthy Eating", and "Exercise") Text messages were positive and motivating and included a link to a specific AADE7 handout that allows participants to open and retrieve the specific AADE7 handout. Text messages were sent by the project investigators to the participants in the intervention group via a free computer-based text messaging service. The computer was password protected and can only be accessed by the investigators. Participant's phone numbers used for text message intervention were kept private. Only investigators and research assistant know the participant's cell phone numbers used for text message intervention and each participant's cell number was not shared with anyone else including other study participants. Text messages were sent by the project investigators or research assistant to the patients and were one-way text messages, meaning that patient did not need to reply to the text messages. If a patient had a medical concern about his/her diabetes, he/she was advised not to send a text message to the investigator, but to contact his/her physician or call 911 instead. The control group did not receive text messages. The participants (both intervention and control group) completed surveys at baseline (before study begins) and at the conclusion of the study (at three month of the intervention) about their dietary and lifestyle habits, diabetes self-care management, awareness of cardiovascular diseases and home food environment. The investigators also collected patient's self-report Hemoglobin A1C values at baseline and at the conclusion of the study (at three month of the intervention).

ELIGIBILITY:
Inclusion Criteria:

* Self-report adult type 2 diabetes patients
* Adults ages 30 or older
* English speaking
* Self-report Hemoglobin A1C > 6.5%
* Have a cell phone able to receive text messages

Exclusion Criteria:

* Individuals without Type 2 diabetes
* Less than 30 years of age
* Self-report Hemoglobin A1C less than 6.5%
* Does not have a cell phone to receive text messages
* Individuals who don't speak and understand English

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Weiwen Chai, PhD, Principal Investigator — University of Nebraska Lincoln
Locations (1):
- University of Nebraska-Lincoln (with Methodist Hospital System), Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cowie CC, Rust KF, Byrd-Holt DD, Gregg EW, Ford ES, Geiss LS, Bainbridge KE, Fradkin JE. Prevalence of diabetes and high risk for diabetes using A1C criteria in the U.S. population in 1988-2006. Diabetes Care. 2010 Mar;33(3):562-8. doi: 10.2337/dc09-1524. Epub 2010 Jan 12. PMID 20067953
- [Background] American Diabetes Association Task Force for Writing Nutrition Principles and Recommendations for the Management of Diabetes and Related Complications. American Diabetes Association position statement: evidence-based nutrition principles and recommendations for the treatment and prevention of diabetes and related complications. J Am Diet Assoc. 2002 Jan;102(1):109-18. doi: 10.1016/s0002-8223(02)90031-3. PMID 11794490
- [Background] Toobert DJ, Hampson SE, Glasgow RE. The summary of diabetes self-care activities measure: results from 7 studies and a revised scale. Diabetes Care. 2000 Jul;23(7):943-50. doi: 10.2337/diacare.23.7.943. PMID 10895844
- [Background] Goodarzi M, Ebrahimzadeh I, Rabi A, Saedipoor B, Jafarabadi MA. Impact of distance education via mobile phone text messaging on knowledge, attitude, practice and self efficacy of patients with type 2 diabetes mellitus in Iran. J Diabetes Metab Disord. 2012 Aug 31;11(1):10. doi: 10.1186/2251-6581-11-10. PMID 23497632
- [Derived] Nepper MJ, McAtee JR, Wheeler L, Chai W. Mobile Phone Text Message Intervention on Diabetes Self-Care Activities, Cardiovascular Disease Risk Awareness, and Food Choices among Type 2 Diabetes Patients. Nutrients. 2019 Jun 11;11(6):1314. doi: 10.3390/nu11061314. PMID 31212683

RESULTS

PARTICIPANT FLOW:
Groups:
- Text Messaging: Participants received 3 messages weekly consisting of nutrition education and diabetes self-management information and skills for 3 months (12 weeks).
  Text messaging: The messages consisted of information on how to increase fruits and vegetables and reduce high-fat and sugary foods intake, increase the availability of fruits and vegetables and reduce high-fat and sugary foods in the home, strategies to increase diabetes self-management skills, and awareness of cardiovascular disease risk perception and knowledge. The text messages will be derived from the American Association of Diabetes Educator (AADE) handouts ("Reducing Risks", "Monitoring", "Healthy Coping", "Problem Solving", "Taking Medication", "Healthy Eating", and "Exercise"). The control group did not receive text messages
- Control: Participants did not receive text message intervention. This is the measurement-only group
Period: Overall Study
Arm/Group | Text Messaging | Control
Started | 40 | 39
Completed | 35 | 35
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Text Messaging: Intervention group received three text messages per week for 12 weeks
- Control: Control group did not receive text messages
- Total: Total of all reporting groups
Arm/Group | Text Messaging | Control | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Customized [Mean (Standard Deviation); unit: years] | 58.8 (10.6) | 55.7 (12.2) | 56.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 14 | 13 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 33 | 36 | 69
  Black | 1 | 2 | 3
  Hispanic | 3 | 0 | 3
  Asian | 1 | 0 | 1
  other | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 39 | 79

OUTCOME MEASURES:

1. Primary Outcome: Self-Care Activities: Healthy Eating
Description: An average of summary scores of the four self-report heathy eating related items in the category (days/over the last 7 days)
Time Frame: Three months
Population: Treatment effects were evaluated by assessing the differences in the outcome variables from baseline to the 12-week follow-up between participants in the intervention group and the control group using Proc Glimmix procedure.
Measure: Least Squares Mean (Standard Error); unit: days/week (min: 0 days; Max: 7 days)
Arm/Group | Text Messaging | Control
Number analyzed (Participants) | 40 | 39
days/week (min: 0 days; Max: 7 days)
  Baseline | 4.23 (0.38) | 4.67 (0.40)
  post-intervention | 4.61 (0.40) | 4.60 (0.41)

2. Primary Outcome: Diabetes Self-care Activity: Exercise
Description: Average of two self-report survey questions related to exercise in the category (days/over the last 7 days)
Time Frame: Three months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days/week (min: 0 days; Max: 7 days)
Arm/Group | Text Messaging | Control
Number analyzed (Participants) | 40 | 39
days/week (min: 0 days; Max: 7 days)
  Baseline | 5.13 (0.62) | 4.91 (0.66)
  post-intervention | 4.48 (0.66) | 4.25 (0.69)

3. Primary Outcome: Self-care Activity: Blood Glucose Testing
Description: Average of two self-report survey question items related to blood glucose testing in the category (days over the last seven days)
Time Frame: three months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days/ week (min: 0 days; max: 7 days))
Arm/Group | Text Messaging | Control
Number analyzed (Participants) | 40 | 39
days/ week (min: 0 days; max: 7 days))
  Baseline | 5.09 (0.64) | 5.93 (0.69)
  post-intervention | 5.27 (0.68) | 5.63 (0.70)

4. Primary Outcome: Self-care Activity: Medication Adherence
Description: Self-report survey question (days over the last seven days)
Time Frame: three months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: day/week (min: 0 days; max 7 days)
Arm/Group | Text Messaging | Control
Number analyzed (Participants) | 40 | 39
day/week (min: 0 days; max 7 days)
  Baseline | 5.75 (0.22) | 5.83 (0.23)
  post-intervention | 5.73 (0.23) | 5.67 (0.24)

5. Primary Outcome: Self-care Activity: Foot Care
Description: Average of four self-report survey questions of the category (days over the last seven days)
Time Frame: three months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: day/week (min: 0 days; max 7 days)
Arm/Group | Text Messaging | Control
Number analyzed (Participants) | 40 | 39
day/week (min: 0 days; max 7 days)
  Baseline | 4.17 (0.41) | 4.22 (0.45)
  post-intervention | 4.89 (0.44) | 4.18 (0.45)

6. Primary Outcome: Eat >= 5 Servings Fruit and Vegetables
Description: Self report survey question (days/week)
Time Frame: Three months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: day/week (min: 0 days; max 7 days)
Arm/Group | Text Messaging | Control
Number analyzed (Participants) | 40 | 39
day/week (min: 0 days; max 7 days) | 4.1 (0.4) | 4.0 (0.3)

7. Secondary Outcome: Self-report Hemoglobin A1C
Description: Self-report hemoglobin for diabetes status
Time Frame: Three months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of glycated HB in blood
Arm/Group | Text Messaging | Control
Number analyzed (Participants) | 40 | 39
percentage of glycated HB in blood
  Baseline | 7.9 (0.3) | 8.5 (0.3)
  post-intervention | 7.6 (0.3) | 8.0 (0.3)

8. Secondary Outcome: Frequency of Concern of CVD Event
Description: Self-report question to measure a patient's cardiovascular disease awareness: Frequency of concern of CVD event
Time Frame: Three months
Population: Chi-square
Measure: Count of Participants; unit: Participants
Arm/Group | Text Messaging | Control
Number analyzed (Participants) | 40 | 39
Participants
  Baseline: Never/rare concern | 28 | 26
  Baseline: Sometimes concern | 9 | 10
  Baseline: Always concern | 3 | 3
  Baseline: Not answer | 0 | 0
  post-intervention: Never/rare concern | 24 | 29
  post-intervention: Sometimes concern | 7 | 5
  post-intervention: Always concern | 4 | 1
  post-intervention: Not answer | 5 | 4

9. Secondary Outcome: Total Carbohydrate
Description: A self-report food frequency questionnaire over the past month
Time Frame: One month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: gram/day
Arm/Group | Text Messaging | Control
Number analyzed (Participants) | 40 | 39
gram/day
  Baseline | 126 (10) | 111 (10)
  post-intervention | 102 (11) | 100 (11)

10. Secondary Outcome: Metabolic Equivalent (MET) Minutes Per Week for Moderate/Vigorous Physical Activity
Description: A Self-report physical activity measure over the past month. The activities were converted to metabolic equivalent (MET: a measure of exercise intensity based on oxygen consumption) minutes per week for moderate/vigorous physical activity
Time Frame: Three months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: MET minutes/week
Arm/Group | Text Messaging | Control
Number analyzed (Participants) | 40 | 39
MET minutes/week
  Baseline | 2112 (1451) | 1042 (1430)
  post-intervention | 3163 (1555) | 405 (1532)

11. Secondary Outcome: Awareness of Cardiovascular Disease (CVD): Degree of Concern of CVD Event in Next 5 Years
Description: Self report survey question
Time Frame: Three months
Population: Chi-square
Measure: Count of Participants; unit: Participants
Arm/Group | Text Messaging | Control
Number analyzed (Participants) | 40 | 39
Participants
  Baseline: No or low concern | 24 | 23
  Baseline: Somewhat concern | 13 | 11
  Baseline: Highly concern | 3 | 5
  Baseline: Not answer | 0 | 0
  post-intervention: No or low concern | 19 | 24
  post-intervention: Somewhat concern | 11 | 8
  post-intervention: Highly concern | 5 | 3
  post-intervention: Not answer | 5 | 4

12. Secondary Outcome: Degree of Concern of CVD Event in Lifetime
Description: Self-report survey question on Cardiovascular disease (CVD) awareness: degree of concern of CVD event in lifetime
Time Frame: Three months
Population: Chi-square
Measure: Count of Participants; unit: Participants
Arm/Group | Text Messaging | Control
Number analyzed (Participants) | 40 | 39
Participants
  Baseline: No concern/low concern | 17 | 12
  Baseline: Somewhat concern | 15 | 20
  Baseline: highly concern | 8 | 7
  Baseline: Not answer | 0 | 0
  post-intervention: No concern/low concern | 12 | 13
  post-intervention: Somewhat concern | 14 | 13
  post-intervention: highly concern | 9 | 9
  post-intervention: Not answer | 5 | 4

ADVERSE EVENTS:
Time Frame: 3 month
Arm/Group | Text Messaging | Control
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 0/40 | 0/39

LIMITATIONS AND CAVEATS:
1) The non-randomized, quasi-experimental study design; 2) Using self-report measures

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT03039569/Prot_SAP_000.pdf